CLINICAL TRIAL: NCT00625521
Title: Efficacy and Safety of ASF-1096 Cream 0.5% in the Treatment of Patients With Newly Developed Discoid Lupus Erythematosus (DLE) Lesions. An International Multi-Centre Clinical Phase 2, Placebo Controlled and Double Blind Proof of Concept Study
Brief Title: Efficacy and Safety of ASF-1096 Cream 0.5% in the Treatment of Discoid Lupus Erythematosus (DLE) Lesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astion Pharma A/S (Industry)
Responsible Party: Dr. Peder M Andersen, Astion Pharma A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASF1096-201
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Discoid Lupus Erythematosus
Keywords: Discoid lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug: ASF 1096 0.5 % cream applied twice daily
  Interventions: Drug: ASF 1096 0.5 % cream applied twice daily
- 2 (Placebo Comparator): Cream vehicle for ASF 1096 cream applied twice daily
  Interventions: Drug: Cream vehicle for ASF 1096 cream applied twice daily

INTERVENTIONS:
Drug: ASF 1096 0.5 % cream applied twice daily
  Arms: 1
Drug: Cream vehicle for ASF 1096 cream applied twice daily
  Arms: 2

SUMMARY:
Lupus Erythematosus (LE) is an autoimmune disorder that includes a broad spectrum of clinical forms. One of these forms, Discoid Lupus Erythematosus (DLE) is a chronic disfiguring disease confined to the skin.

The aim of this pivotal trial is to investigate the efficacy and safety of ASF-1096 cream 0.5% in the treatment of patients with DLE or SLE presenting newly developed discoid lesions.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of either DLE or SLE
* Histological results from biopsy confirming the diagnosis (biopsy can be taken at screening)
* Is prepared to grant authorised persons access to the medical records
* Has signed informed consent

Exclusion Criteria:

* Has an active skin disease other than DLE or another progressive or serious disease that interferes with the study outcome
* Has scarring at the target lesion
* Systemic treatment of SLE

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-11; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety profile, CLASI score, GIA and GPA.

CONTACTS AND LOCATIONS:
Locations (1):
- Filippa Nyberg, Danderyd Stockholm, Sweden